CLINICAL TRIAL: NCT05875415
Title: Dynamic Plantar Pressures Changes After Dry Needling in Flexor Digitorum Brevis Versus Non Emission Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist., Mayuben Private Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1912202200923-B
Record Dates: First submitted 2023-05-15; First posted 2023-05-25 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Flatfoot
Keywords: Foot; gait; Dry Needling; trigger point
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral dry needling in Flexor Brevis Digitorum in subjects with latent trigger point (Experimental)
  Interventions: Other: Bilateral dry needling in latent trigger points of the Flexor digitorum Brevis Muscle
- Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle (Sham Comparator)
  Interventions: Other: Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle

INTERVENTIONS:
Other: Bilateral dry needling in latent trigger points of the Flexor digitorum Brevis Muscle — Bilateral dry needling in latent trigger points of the Flexor digitorum Brevis Muscle in flatfoot
  Arms: Bilateral dry needling in Flexor Brevis Digitorum in subjects with latent trigger point
Other: Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle — Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle in flatfoot
  Arms: Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle

SUMMARY:
Thirty-six subjects randomly distributed between a dry needling intervention group and a control group whose intervention is a non-emission laser. All the subjects will be measured before and after the interventions of each group. The measurements will be made on a pressure platform to record the dynamic footprint variables.

DETAILED DESCRIPTION:
Thirty-six subjects randomly distributed between a dry needling intervention group and a control group whose intervention is a non-emission laser. All the subjects will be measured before and after the interventions of each group. The measurements will be made on a pressure platform to record the dynamic footprint variables of the first step of both feet.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have latent trigger point in Flexor Brevis Digitorum muscles with no other pathologies

Exclusion Criteria:

* Previous lower extremities surgery.
* History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.
* Leg-length discrepancy more than 1 cm
* Balance deficits (determined by oral questionnaire regarding falls)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Surface before dry needling in right foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface before dry needling in right foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2)
Surface before dry needling in right foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface before dry needling in right foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)
Surface before dry needling in left foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface before dry needling in left foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2)
Surface before dry needling in left foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface before dry needling in left foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)
Surface after dry needling in right foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface after dry needling in right foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2)
Surface after dry needling in right foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface after dry needling in right foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)
Surface after dry needling in left foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface after dry needling in left foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2)
Surface after dry needling in left foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface after dry needling in left foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)
Surface before Laser non-emission in right foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface before Laser non-emission in right foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2).
Surface before Laser non-emission in right foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface before Laser non-emission in right foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)
Surface before Laser non-emission in left foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface before Laser non-emission in left foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2).
Surface before Laser non-emission in left foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface before Laser non-emission in left foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)
Surface after Laser non-emission in right foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface after Laser non-emission in right foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2).
Surface after Laser non-emission in right foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface after Laser non-emission in right foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)
Surface after Laser non-emission in left foot at 20% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 20% of the total duration, measured in square centimeters (cm2)
Surface after Laser non-emission in left foot at 35% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 35% of the total duration, measured in square centimeters (cm2).
Surface after Laser non-emission in left foot at 92% of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the dynamic footprint at 92% of the total duration, measured in square centimeters (cm2)
Surface after Laser non-emission in left foot at Global of time of first step | Through study completion, an average of 1 week
  Registration of the surface of the global dynamic footprint of the total duration, measured in square centimeters (cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Eva María MartínezJiménez, Principal Investigator — Mayuben Clinic
Locations (1):
- Eva María Martínez-Jimenez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No